CLINICAL TRIAL: NCT05430750
Title: Global Warming Impact and Clinical Effects of a Novel 'streamed-in' Nitrous Oxide Administration as a Carrier Gas During Sevoflurane General Anaesthesia: a Randomized Pilot Study
Brief Title: Global Warming Impact of Nitrous Oxide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Associate Professor & Senior Consultant, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EC/05/22/2063
Record Dates: First submitted 2022-06-18; First posted 2022-06-24 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Global Warming Effect of Nitrous Oxide
Keywords: nitrous oxide; sevoflurane; global warming
MeSH Terms: interventions — Nitrous Oxide; Sevoflurane

STUDY DESIGN:
Intervention Model Description: One hundred and two patients of either sex, and schedule for elective surgery under general anesthesia (GA) will be randomly divided into three groups of 34-each.
  Group 1('Conventional' N2O carrier gas group) Ventilation will be initiated with 2% Sevoflurane in O2-N2O (60 % FiO2) @3L/min to MAC 0.5. Once MAC reaches 0.5, the FGF will be decreased to 1.0L/min.
  Group 2 ('Streamed-in' N2O carrier gas group) Ventilation will be initiated with 2% Sevoflurane in O2 -Air (60 % FiO2) @3.0L/min to achieve a MAC of 0.5. Then, the FGF will be decreased to 1.0 L (low flow) and N2O will be 'streamed-in' @ 40 %.
  Group 3 (Non-N2O group) Ventilation will be initiated with 2% Sevoflurane in O2-Air (60 % FiO2 @ 3.0L/min) till the time it reaches MAC 0.5. Once MAC 0.5 reached, the FGF is decreased to 1.0L (Low-flow).
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to the type of anesthesia intervention. The attending anesthesiologist will however not be blinded to the technique utilized to administer GA and recovery immediately after extubation inside the OR. The postoperative patient profile will be evaluated by an independent assessor blinded to the technique of GA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional' - N2O carrier gas group (Active Comparator): Ventilation will be initiated with 2% Sevoflurane in O2-N2O (60 % FiO2) @3L/min to MAC 0.5. Once MAC reaches 0.5, the FGF will be decreased to 1.0L/min (Low flow) and allowed to reach MAC 1.0 before incision is allowed. At 20-minutes time point post induction if MAC 1.0 is not achieved at 2% sevoflurane then the sevoflurane vaporizer concentration will be adjusted to achieve MAC 1.0, before incision is allowed. Anaesthesia will be maintained at MAC 1.0 throughout. After surgery is over, the N2O - Sevoflurane will be stopped and FGF increased to 3.0L with 100% O2.
  Interventions: Drug: Nitrous oxide; Drug: Sevoflurane
- 'Streamed -in' N2O carrier gas group (Active Comparator): Ventilation will be initiated with 2% Sevoflurane in O2 -Air (60 % FiO2) @3.0L/min to achieve a MAC of 0.5. Then, the FGF will be decreased to 1.0 L (low flow) and N2O will be 'streamed-in' @ 40 %. When MAC 1.0 is reached incision will be allowed. At 20-minutes time point post induction if MAC 1.0 is not achieved at 2% sevoflurane then the sevoflurane vaporizer concentration will be adjusted to achieve MAC 1.0, before incision is allowed. Anaesthesia will be maintained at MAC 1.0 throughout. After surgery is over, the N2O - Sevoflurane will be stopped and FGF increased to 3.0L with 100% O2.
  Interventions: Drug: Nitrous oxide; Drug: Sevoflurane
- Non-N2O group (Active Comparator): Ventilation will be initiated with 2% Sevoflurane in O2-Air (60 % FiO2 @ 3.0L/min) till the time it reaches MAC 0.5. Once MAC 0.5 reached, the FGF is decreased to 1.0L (Low-flow). The incision is allowed when MAC 1.0 is achieved .At 20-minutes time point post induction if MAC 1.0 is not achieved at 2% sevoflurane then the sevoflurane vaporizer concentration will be adjusted to achieve MAC 1.0, before incision is allowed. Anaesthesia will be maintained at MAC 1.0 throughout. After surgery is over, the O2 - Sevoflurane will be stopped and FGF increased to 3.0L with 100% O2.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Nitrous oxide — In conventional nitrous oxide carrier group 2% Sevoflurane in O2-N2O (60 % FiO2) @3L/min will be delivered to achieve MAC 0.5.
  Arms: Conventional' - N2O carrier gas group
Drug: Nitrous oxide — In streamed-in nitrous oxide carrier group 2% Sevoflurane in O2 -Air (60 % FiO2) will be delivered @3.0L/min to achieve a MAC of 0.5. Then, the FGF will be decreased to 1.0 L (low flow) and N2O will be 'streamed-in' @ 40 %.
  Arms: 'Streamed -in' N2O carrier gas group
Drug: Sevoflurane — Ventilation will be initiated with 2% sevoflurane in all the groups

SUMMARY:
Environmental hazards of human activity are a topic of present day world, global warming being one of the leading concerns. Gases that contribute to this are greenhouse gases. Nitrous oxide (N2O) is a greenhouse gas that is commonly used in medical practice, mostly confined to provision of anaesthesia during surgical procedures in the operation theatre. N2O is not a potent anesthetic, and is used as a carrier for volatile anesthetic during general anaesthesia. This is to reduce the use of volatile anesthetics and other analgesic drugs while maintaining adequate depth of anaesthesia and analgesia. The N2O gas that is used during general anaesthesia is scavenged and released into the atmosphere without any processing. In the atmosphere it stays and produces deleterious greenhouse effect primarily owing to its long lifetime of 114 years. In addition, it also causes depletion of ozone layer. The green house effect of gases is evaluated and compared with the use of carbon-di-oxide equivalents (CDE). When the effects are considered for 20 years it is termed CDE20.The efforts to reduce these harmful effects can be directed towards reduction/cessation of N2O use, or its post anesthetic processing. The long history of its use in clinical practice and benefits such as analgesia for various procedures; makes it difficult to be completely taken out of usage in the present day anaesthesia practice. Though processing of N2O after use during GA is possible, it's impractical because of cost efficiency. We therefore, have directed our focus on further reducing its consumption while being used for GA. Low- flow anaesthesia has been in practice for the same reason (i.e. to reduce the wastage of gases).

This study is aimed to reduce the N2O consumption even further by employing a novel 'streamed-in' technique of N2O administration during low-flow GA. Conventionally, N2O use is initiated during the initial high fresh gas flows (FGF) before shifting to low-flow ventilation. 'Streamed-in' N2O administration strategy employs initiation of N2O into FGF after the institution of low-flow anaesthesia. Hence, the participants are not exposed to an unconventional drug or a new route of its administration, but an alternate strategy to its conventional use. We aim to evaluate the novel technique of 'streamed-in' N2O during sevoflurane GA for its global warming effects (in terms of CDE20) and its clinical effects ( intraoperative general anaesthesia state, hemodynamic profile) and post operative effects( postoperative nausea vomiting -PONV, postoperative pain profile- numerical rating scale-NRS)

DETAILED DESCRIPTION:
Earliest use of nitrous oxide (N2O) in medical practice dates back to 1884. It aimed at providing analgesia during surgical procedure. Over the years the N2O use for anaesthesia evolved with the knowledge that it has very low anesthetic potential and high minimum alveolar concentration (MAC =104%), and therefore it cannot be used as a sole anesthetic. This led to N2O being used a carrier gas only during inhalational vapor (sevoflurane, isoflurane, desflurane) anaesthesia. The N2O- vapor co-administration not only reduces inhaled vapor requirements but also offers continuous analgesia state during maintenance of anaesthesia. Studies show its use in sedation and analgesia for labor analgesia and other minor procedures especially in pediatric population, such as, venipuncture, venous cannulation, fracture reduction, lumbar puncture, acute pain etc. Further, the use of intraoperative N2O also reduces the incidence of patients developing chronic postoperative pain.

The use of N2O, with attendant application advantages come the disadvantages of having undesirable effect on the patient (diffusion hypoxia, PONV), the medical care provider (megaloblastic anemia, risk of spontaneous abortion, reduced fertility) and environment (global warming). N2O possesses greenhouse effect defined in terms of global warming potential (GWP) [20 year GWP and 100year GWP - 289 (GWP20) and 298 (GWP100), respectively] and 'ozone depleting' properties. The above stated effects in conjunction with long life-span of N2O (114 years) in the atmosphere is likely to lead to longstanding negative environmental impact if its use is not stopped/made more efficient. Therefore, there is an absolute need for using N2O more efficiently for reducing effects on the patients, the first to get exposed operative room personnel, and ambient environment at large.

Sevoflurane is an inhalational anesthetic with a sweet smell, fast onset, offset and a good safety profile. Sevoflurane is also a greenhouse gas. Its use in combination with N2O is in practice for the benefits discussed earlier.

Having been in medical use for over 150 years with its various benefits, the use of N2O cannot be expected to be abandoned in the near future. Though steps to reduce anesthetic gas usage with techniques such as low-flow anaesthesia (fresh gas flow-FGF<alveolar ventilation, arbitrarily taken as 2L/min) and safer carbon-di-oxide absorbers are in vogue; no further/specific exploration has been undertaken. With Sevoflurane, use of fresh gas flows less than 1L/min is not recommended due to concerns surrounding production of Compound A and its nephrotoxic effects (clinically unproven in human ).

Inhalational anesthetics are almost completely excreted through lungs via exhalation without undergoing significant metabolism. Even ex-vivo inhalational agents are not processed, but only collected through scavenging system and released into the atmosphere. 15 The use of N2O with inhalational anesthetics leaves a far greater impact on the environment when compared to their use with air/O2. Though N2O's pound-for- pound impact in terms of global warming (GWP20-289) is less when compared to other inhalational anesthetics in use [ isoflurane (GWP20-1401), sevoflurane (GWP20-349), desflurane (GWP20-3714)]; it has a more significant impact on environment mainly because of the much higher consumption volume and also the fact that it is a 'stock' pollutant i.e. has a long lifetime and accumulates overtime. In contrast, inhalational anesthetics which are 'flow' pollutants i.e. have short lifetime and doesn't accumulate as long as new release into atmosphere is kept constant. The global warming impact of gases is evaluated and compared by the CO2 equivalents (CDE) produced. CDE20 (Anesthetic gas quantity in grams *GWP20), takes into account both the GWP and the quantity of the gas that is produced. The GWP and CDE are calculated for a defined duration of time. Commonly implemented in case of inhalational anesthetic is for 20 years, as the atmospheric lifetime of inhalational anesthetics is less than 20 years.

With the growing concern for global warming and impact of human activity on the earth's ecology; medical fraternity should be at the forefront of new developments that work towards these issues. With the subject at hand the investigators are attempting to reduce the medical use of N2O and in turn its effects on the environment by evaluating a novel method of N2O use. We expect it to reduce the N2O consumption significantly enough to lessen its harmful global ecological impact.

Conventional low-flow anaesthesia with N2O is implemented by using FGF of about ≥4L/m (O2 + N2O) initially. Once desired anesthetic gas composition is attained in the system and the minimum alveolar concentration reflects adequacy of anesthetic depth (i.e. MAC 0.7-1.3), FGF is reduced to the low-flow i.e. ≤1.0 Liters/min.

Though there is evidence to negative environmental effects of inhaled anesthetic vapor and N2O, they have been largely based on theoretical methodology. To the best of our knowledge, till date there are no studies that have evaluated the global warming effects of inhaled GA (with and without N2O) on real use-in patient scenarios. Given that different patients may have different anesthetic uptake (N2O, inhaled vapor) characteristics with different strategies of GA, the consequent environmental effect may be variable, and therefore, must be quantified and controlled.

In this proposed study, the investigators aim to evaluate a novel technique of N2O administration i.e. "streamed-in" administration technique in terms of its global warming impact and clinical effects. Initially, air-O2-sevoflurane is introduced at high FGF of 3.0 L/min. Once the target anesthetic gas concentration is attained in the system i.e. MAC 0.5, FGF is reduced to achieve a low-flow state. At this point N2O is "streamed-in" to add to O2-sevoflurane mixture.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA physical status I and II
* Patients undergoing elective non-laparoscopic surgeries of minimum 1 hour duration without use of adjuvant central neuraxial or peripheral nerve block under general anaesthesia

Exclusion Criteria:

* Failure to obtain consent
* Neurological disorders (previous neurosurgery , psychiatric disorders, autonomic system disorders - orthostatic hypotension, transient ischemic attacks )
* Cardiovascular disorders (uncontrolled hypertension, A-V block, sinus bradycardia, congenital heart disease, reduced LV compliance and diastolic dysfunction)
* Hepatorenal insufficiency
* Uncontrolled endocrine disorders (diabetes mellitus, hypothyroidism, hyperthyroidism)
* Electrolyte disturbances (hyponatremia, hypernatremia)
* Pulmonary dysfunction (restrictive /obstructive lung disease)
* Acute /chronic drug dependence /substance abuse
* Closed cavity surgeries (middle ear surgeries, eye surgeries)
* Previous h/o PONV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Carbon-di-oxide equivalent -20 years (CDE20) | From start of anesthesia till 5- minutes post extubation
  Carbon-di-oxide equivalent -20 years of nitrous oxide & sevoflurane will be calculated using the formula Mass of Anaesthetic used *GWP20 (Global Warming Potential -20 years)

SECONDARY OUTCOMES:
Intraoperative End-tidal anaesthesia gas (ETAG) concentration | From start of anesthesia till 5- minutes post extubation
  ETAG concentration of nitrous oxide, sevoflurane, oxygen, carbon dioxide will be recorded from the patient monitor
Intraoperative minimum alveolar concentration (MAC) | From start of anesthesia till 5- minutes post extubation
  MAC will be recorded from the patient monitor
Intraoperative consumption of anesthetic gases | From start of anesthesia till 5- minutes post extubation
  Intraoperative consumption of nitrous oxide, sevoflurane, oxygen and air will be noted at the end of anesthesia from the log book of the anesthesia machine
Changes in intra-operative heart rate (beats per minute) | From start of anesthesia till 5- minutes post extubation
  Comparison of intra-operative heart rate will be done among the three groups
Change in Intra-operative blood pressure - systolic , diastolic, and mean (mmHg) | From start of anesthesia till 5- minutes post extubation
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean will be done among the three groups
Changes in rate pressure product | From start of anesthesia till 5- minutes post extubation
  Comparison of rate pressure product will be done among the three groups. Rate pressure product will be calculated using the formula :Systolic blood pressure *heart rate /1000
Postoperative Nausea and Vomiting (PONV) | From end of anaesthesia till 24-hours postoperatively
  PONV will be assessed using postoperative nausea and vomiting (PONV) Scale. The scale measures PONV on a scale of 0 to 2. A score of '0' indicates that the patient has no emetic symptoms, whereas a score of '2' indicates that the patient has vomiting.
Postoperative pain | From end of anaesthesia till 24-hours postoperatively
  Postoperative pain will be assessed using the 10-point numerical rating scale. The scale has scoring from 0 to 10. '0' implying minimum pain & '10' implying maximum pain
Incidence of intraoperative awareness | From end of anaesthesia till 24-hours postoperatively
  Awareness will be assessed using 5-question based Brice Structured Interview

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Dutta, MD, PGDHR, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Nitin Sethi, DNB, Study Director — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No